CLINICAL TRIAL: NCT04097938
Title: A First-in-human Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Oral Doses of GLPG3667 in Adult, Healthy, Male Subjects
Brief Title: A Study to Evaluate the Effects of Single and Multiple Oral Doses of GLPG3667
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galapagos NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: GLPG3667-CL-101; 2019-001659-38 (EudraCT Number)
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2020-07

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (9):
- GLPG3667 SAD (Experimental): Single doses of GLPG3667 at up to 6 dose levels in ascending order
  Interventions: Drug: GLPG3667 oral suspension
- Placebo SAD (Placebo Comparator): Single doses of placebo
  Interventions: Drug: Placebos
- GLPG3667 MAD (Experimental): Multiple doses of GLPG3667 at up to 3 dose levels in ascending order, daily for 13 days
  Interventions: Drug: GLPG3667 oral suspension
- Placebo MAD (Placebo Comparator): Multiple doses of placebo
  Interventions: Drug: Placebos
- GLPG3667 FE fasted (Experimental): Single dose of GLPG3667 in fasted state
  Interventions: Drug: GLPG3667 oral suspension
- GLPG3667 FE fed (Experimental): Single dose of GLPG3667 in fed state
  Interventions: Drug: GLPG3667 oral suspension
- GLPG3667 oral suspension rBA-FE fed (Experimental): Single dose of GLPG3667 oral suspension in fed state
  Interventions: Drug: GLPG3667 oral suspension
- GLPG3667 capsules rBA-FE fasted (Experimental): Single dose of GLPG3667 capsules in fasted state
  Interventions: Drug: GLPG3667 capsules
- GLPG3667 capsules rBA-FE fed (Experimental): Single dose of GLPG3667 capsules in fed state
  Interventions: Drug: GLPG3667 capsules

INTERVENTIONS:
Drug: GLPG3667 oral suspension — GLPG3667 oral suspension
  Arms: GLPG3667 FE fasted; GLPG3667 FE fed; GLPG3667 MAD; GLPG3667 SAD; GLPG3667 oral suspension rBA-FE fed
Drug: Placebos — Placebo oral suspension
  Arms: Placebo MAD; Placebo SAD
Drug: GLPG3667 capsules — GLPG3667 capsules
  Arms: GLPG3667 capsules rBA-FE fasted; GLPG3667 capsules rBA-FE fed

SUMMARY:
This study is a first-in-human, Phase I, randomized, double-blind, placebo-controlled, single-center, dose-escalation study to evaluate the safety, tolerability, pharmacokinetics (PK) and pharmacodynamics of GLPG3667 after oral single ascending doses (SAD) of GLPG3667 (part 1) and after oral multiple ascending doses (MAD) for 13 days of GLPG3667 (part 2) in healthy male subjects. In addition, the effect of food (FE) on safety, tolerability, and PK of GLPG3667 oral suspension will be evaluated (part 3 - will not be completed), and the relative bioavailability (rBA) of the capsule versus the oral suspension with the effect of food on the bioavailability of the capsule (part 4), both part 3 and 4 using an open-label, randomized, crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Male between 18-55 years of age (extremes included), on the date of signing the informed consent form (ICF)
* A body mass index (BMI) between 18-30 kg/m2, inclusive
* Judged to be in good health by the investigator based upon the results of a medical history, physical examination, vital signs, 12-lead electrocardiogram (ECG), and fasting clinical laboratory safety tests, available at screening and prior to randomization. Hemoglobin, neutrophil, lymphocyte, and platelet counts must be above the lower limit of normal range. Bilirubin, aspartate aminotransferase (AST), and alanine aminotransferase (ALT) must be within normal ranges. Other clinical laboratory safety test results must be within the reference ranges or test results that are outside the reference ranges need to be considered not clinically significant in the opinion of the investigator

Exclusion Criteria:

* Known hypersensitivity to Investigational Medicinal Product (IMP) ingredients or history of a significant allergic reaction to IMP ingredients as determined by the investigator
* Known contraindication or hypersensitivity to Interferon-alpha (IFN-α) or any component of Intron-A® (Note: this criterion is only applicable to subjects in the MAD part)
* Positive serology for hepatitis B virus surface antigen (HBsAg) or hepatitis C virus (HCV) or history of hepatitis from any cause with the exception of hepatitis A that was resolved at least 3 months prior to first dosing of the IMP.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2019-09-18 (Actual); Primary Completion 2020-03-04 (Actual); Study Completion 2020-07-06 (Actual)

PRIMARY OUTCOMES:
Frequency and severity of treatment-emergent adverse events (TEAEs), treatment-emergent serious adverse events, and TEAEs leading to treatment discontinuations | From screening through study completion, an average of 5 months
  To evaluate the safety and tolerability of single and multiple ascending oral doses of GLPG3667, in adult, healthy, male subjects compared with placebo

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of GLPG3667 (μg/mL) | Between Day 1 pre-dose and Day 16
  To evaluate the pharmacokinetics (PK) of single and multiple ascending oral doses of GLPG3667, in adult, healthy, male subjects
Area under curve (AUC) of GLPG3667 (μg.h/mL) | Between Day 1 pre-dose and Day 16
  To evaluate the PK of single and multiple ascending oral doses of GLPG3667, in adult, healthy, male subjects
Terminal elimination half-life (t1/2) of GLPG3667 (h) | Between Day 1 pre-dose and Day 16
  To evaluate the PK of single and multiple ascending oral doses of GLPG3667, in adult, healthy, male subjects

CONTACTS AND LOCATIONS:
Overall Officials: Magdalena Petkova, MD, Study Director — Galapagos NV
Locations (1):
- SGS Belgium NV - Clinical Pharmacology Unit Antwerp, Antwerp, Belgium

IPD SHARING:
Plan to Share IPD: No